CLINICAL TRIAL: NCT05080998
Title: An Observational Study of CxBladder Monitoring for Recurrence of Urothelial Carcinoma in Low-, Intermediate-, and High-Risk Patients
Brief Title: Longitudinal Bladder Cancer Study for Tumour Recurrence
Acronym: LOBSTER
Status: Recruiting | Type: Observational
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CXBM/2021/VA
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Bladder Cancer
Keywords: Recurrence
MeSH Terms: conditions — Recurrence | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and tissue specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm - Patients undergoing surveillance for UC recurrence: Subjects previously diagnosed with UC and are undergoing a schedule of surveillance cystoscopies and treatment for the possible recurrence of UC will be recruited. Low-, intermediate-, and high-risk groups, according to AUA /SUO risk categorisation for non-muscle invasive UC, will be eligible for this study. All subjects will undergo CxBladder urine diagnostic testing.
  Interventions: Diagnostic Test: CxBladder Monitor/Monitor+

INTERVENTIONS:
Diagnostic Test: CxBladder Monitor/Monitor+ — CxBladder Monitor/Monitor+ is a high sensitivity and negative predictive value (NPV) urinary biomarker test to rule-out subjects at low risk of bladder cancer monitoring for recurrence of disease.

SUMMARY:
Surveillance for recurrence of urothelial carcinoma (UC) requires frequent cystoscopy, which is invasive, expensive and time-consuming. An accurate urinary biomarker has the potential to reduce the number of cystoscopies required during post-treatment surveillance. This is a prospective, single arm, multi-center study using the diagnostic CxBladder test with subjects previously diagnosed with primary or recurrent UC and who are undergoing a schedule of investigative cystoscopies and treatment for the possible recurrence of UC presenting to qualified sites. To evaluate the performance characteristics of the CxBladder test, multiple consecutive urine samples will be collected during the course of surveillance.

DETAILED DESCRIPTION:
This is a multi-site study recruiting subjects from Veterans Affairs and other medical centers. Subjects will be prospectively recruited to an observational study to validate the performance characteristics of CxBladder Monitor test (Monitor) and the second-generation test, CxBladder Monitor Plus (Monitor+). The study will recruit low, intermediate, and high-risk surveillance subjects, defined as per American Urological Association (AUA) / Society of Urologic Oncology (SUO) guidelines 2016 amendment 2020, previously diagnosed with urothelial carcinoma (UC). Eligible subjects will include those under surveillance for recurrence of UC. A voided urine sample will be collected from each enrolled subject at each of 4 successive surveillance visits. The collected urine will be used for CxBladder testing and central urine cytology. The study will collect primary tumour tissue from the first confirmed tumour, i.e., the primary diagnosis of UC (if available) and any subsequent collections within 12 weeks. Tissue samples from any UC recurrences while in study will also be collected to genotype each tumour using RNA or DNA markers indicative of an elevated risk of UC. Monitor/Monitor+ results will not be reported to patients or physicians. This study primarily aims to clinically validate the performance characteristics (sensitivity, specificity, negative predictive value, positive predictive value, and test-negative rate) of the Cxbladder Monitor/Monitor+ test compared to the reference standard i.e., tumours observed by cystoscopy and confirmed by pathology over a maximum of 4 surveillance visits. Sites are required to be competent in recruiting and completing required test request forms, Case Report Forms (CRF) and sample collection in a professional manner in accordance with good clinical practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

1. Low-, intermediate-, and high-risk surveillance subjects with a previous confirmed diagnosis or recurrence of urothelial carcinoma within the last 3 calendar years.
2. Subjects must agree to 4 successive study visits, including urine sample collection at each visit.
3. Physically able to provide a voided urine sample (a sample from catheterization is not eligible).
4. Able to give written informed consent
5. Able and willing to comply with study requirements
6. Aged 18 years or older

Exclusion Criteria:

1. Total cystectomy of the bladder, subjects with neo-bladders or illeal conduits
2. Previous muscle invasive bladder tumour (pT2 or greater)
3. Known pregnancy

Deferral Criteria

1. Prior genitourinary manipulation (catheterisation, urethral dilation, cystoscopy, etc.) within 14 calendar days of the scheduled urine collection, study enrollment with urine sample collection for Cxbladder Monitor testing should be deferred until a minimum of 14 calendar days has passed since the procedure was performed.
2. Active urinary tract infection (UTI) within 14 calendar days of the scheduled urine collection, study enrollment with urine sample collection for Cxbladder Monitor testing should be deferred until the treatment is complete and the UTI is resolved.
3. If a subject has had intravesical immunotherapy or chemotherapy within the previous 6 weeks, study enrollment with urine sample collection for Cxbladder Monitor testing should be deferred. Study enrollment must be at least 28 calendar days post-last treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit low-, intermediate-, and high-risk surveillance subjects (defined as per AUA/SUP Guidelines 2016, amendment 2020), previously diagnosed with urothelial carcinoma.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To clinically validate the performance characteristics of CxBladder Monitor/Monitor+ | 12 Months
  To clinically validate the performance characteristics - sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV), and test-negative rate of Monitor and Monitor+ for the detection of recurrent UC in subjects with a recent history of urinary tract UC who are being treated according to standard of care and are concurrently undergoing routine investigative cystoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lough, Study Chair — Pacific Edge Pty Ltd
Locations (7):
- United States (6):
  - Miami VA Healthcare System, Miami, Florida
  - James A. Haley Veteran's Hospital, Tampa, Florida
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - White River Junction Veterans Affair Medical Center, White River Junction, Vermont
  - University of Washington School of Medicine, Seattle, Washington
- Monash Health - Moorabbin Hospital, Clayton, Victoria, Australia